CLINICAL TRIAL: NCT00084890
Title: Weekly Docetaxel and Carboplatin in Patients With Recurrent Squamous Carcinoma of the Cervix: A Phase I/II Study
Brief Title: Docetaxel and Carboplatin in Treating Patients With Recurrent Stage IVB Squamous Cell Carcinoma (Cancer) of the Cervix
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000366942; CCCWFU-30102B; NCI-6949
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: stage IVB cervical cancer; recurrent cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: carboplatin — 30 minute infusion dosed based on glomerular filtration rate of patient
Drug: docetaxel — escalating doses ofstarting at 25 milligrams per meter squared

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining docetaxel with carboplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel when given together with carboplatin and to see how well they work in treating patients with recurrent stage IVB squamous cell carcinoma (cancer) of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of docetaxel when administered with carboplatin in patients with recurrent stage IVB squamous cell carcinoma of the cervix.
* Determine the response rate and time to progression in patients treated with this regimen.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is phase I, dose-escalation study of docetaxel followed by a phase II study.

* Phase I: Patients receive docetaxel IV over 30 minutes and carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients who demonstrate continuing tumor shrinkage after 6 courses receive 2 additional courses beyond their best response.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive docetaxel and carboplatin as in phase I at the MTD determined in phase I.

Quality of life is assessed at baseline, before every other course of treatment, and at the end of study treatment.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 3-64 patients (3-24 for phase I and 16-40 for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the uterine cervix

  * Advanced disease (stage IVB)
  * Persistent or recurrent disease
* No available curative treatment options
* Measurable disease by physical examination, chest x-ray, CT scan, or MRI

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* GOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8 g/dL

Hepatic

* Bilirubin normal
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN) AND alkaline phosphatase normal OR
* Alkaline phosphatase ≤ 4 times ULN AND SGOT and SGPT normal

Renal

* Creatinine < 1.5 times ULN

Other

* No other invasive malignancy within the past 5 years
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy > grade 1
* No other concurrent malignancy except curatively treated non-melanoma skin cancer
* No other serious medical or psychiatric illness that would preclude giving informed consent or limit survival
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* No more than 2 prior chemotherapy regimens

  * One sensitizing chemotherapy regimen during radiotherapy AND 1 regimen for recurrent disease are considered 2 regimens
* At least 4 weeks since prior chemotherapy
* No prior docetaxel
* No prior carboplatin
* No other concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior hormonal therapy

Radiotherapy

* See Chemotherapy
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior major surgery

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2007-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of docetaxel | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte E. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States